CLINICAL TRIAL: NCT04383665
Title: Evaluation of Neurocognitive Changes in Parkinson's Disease Patients Following Acute Low Frequency Deep Brain Stimulation
Brief Title: Low Frequency Subthalamic Nucleus Deep Brain Stimulation to Improve Verbal Fluency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Darrin J Lee, MD, PhD, Assistant Professor of Neurosurgery, University of Southern California
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: HS-19-00518
Record Dates: First submitted 2020-05-07; First posted 2020-05-12 (Actual); Results first posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-06

CONDITIONS: Parkinson Disease
Keywords: Cognition; Hippocampus; Language; Memory; Neuromodulation; Randomized controlled trial
MeSH Terms: conditions — Parkinson Disease; Language

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- STN DBS off (Sham Comparator)
  Interventions: Device: STN DBS off
- STN DBS 10Hz (Experimental)
  Interventions: Device: STN DBS 10Hz
- STN DBS 130Hz (Active Comparator)
  Interventions: Device: STN DBS 130Hz

INTERVENTIONS:
Device: STN DBS 10Hz — Stimulation of existing DBS device at 100Hz, with other parameters at baseline
  Arms: STN DBS 10Hz
Device: STN DBS 130Hz — Stimulation of existing DBS device at 130Hz, with other parameters at baseline
  Arms: STN DBS 130Hz
Device: STN DBS off — Existing DBS device turned off
  Arms: STN DBS off

SUMMARY:
Rationale: Parkinson's disease patients with deep brain stimulation electrodes represent a unique opportunity to study the influence of basal ganglia on neurocognitive function.

Intervention: Patients' deep brain stimulators will be turned off or on and the frequency will be changed to either theta or gamma.

Objectives: To identify differences in higher cognitive functions with stimulation "on" and "off" and theta versus gamma frequency stimulation.

Study population: 12 patients who had previously undergone bilateral STN deep brain stimulation implantation.

Study methodology: Patients will undergo four sessions of neuropsychological testing (RNGT, verbal fluency, D-KEFS CWIT) at baseline, no stimulation, theta stimulation and gamma stimulation, in random order over one day.

Study outcomes: Test results of RNGT, verbal fluency, D-KEFS CWIT. Follow-up: none

Statistics: Test results will be analyzed using within-subjects statistical tests.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients who had previously undergone bilateral STN deep brain stimulation implantation
2. Age >18 years old
3. Stable medication regimen for at least 3 months.
4. Patient informed and able to give written consent
5. Able to comply with all testing, follow-ups and study appointments and protocols

Exclusion Criteria:

1. History of epilepsy or seizure
2. History of major substance abuse
3. Patients with baseline settings at less than 1.5 V will be excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2020-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darrin J Lee, MD PhD, Principal Investigator — University of Southern California
Locations (1):
- Keck hospital of the University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Evans FJ. Monitoring attention deployment by random number generation: An index to measure subjective randomness. Bull Psychon Soc 1978;12:35-8.
- [Background] Spatt J, Goldenberg G. Components of random generation by normal subjects and patients with dysexecutive syndrome. Brain Cogn. 1993 Nov;23(2):231-42. doi: 10.1006/brcg.1993.1057. PMID 8292327
- [Background] Towse JN, Neil D. Analyzing human random generation behavior: A review of methods used and a computer program for describing performance. Behav Res Methods Instrum Comput 1998;30:583-91.
- See also: RGCalc — https://www.lancaster.ac.uk/staff/towse/rgcpage.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 12 participants, each tested at off, 10 Hz and 130 Hz
Groups:
- Off/10 Hz/130 Hz: 1. STN DBS device turned off
  2. STN DBS at 10 Hz
  3. STN DBS at 130 Hz
- Off/130 Hz/10 Hz: 1. STN DBS device turned off
  2. STN DBS at 130 Hz
  3. STN DBS at 10 Hz
- 10 Hz/Off/130 Hz: 1. STN DBS at 10 Hz
  2. STN DBS device turned off
  3. STN DBS at 130 Hz
- 10 Hz/130 Hz/Off: 1. STN DBS at 10 Hz
  2. STN DBS at 130 Hz
  3. STN DBS device turned off
- 130 Hz/Off/10 Hz: 1. STN DBS at 130 Hz
  2. STN DBS device turned off
  3. STN DBS at 10 Hz
- 130 Hz/10 Hz/Off: 1. STN DBS at 130 Hz
  2. STN DBS at 10 Hz
  3. STN DBS device turned off
Period: Overall Study
Arm/Group | Off/10 Hz/130 Hz | Off/130 Hz/10 Hz | 10 Hz/Off/130 Hz | 10 Hz/130 Hz/Off | 130 Hz/Off/10 Hz | 130 Hz/10 Hz/Off
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All Study Participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 12
Primary language [Count of Participants; unit: Participants]
  English | 9
  Spanish | 2
  Chinese | 1

OUTCOME MEASURES:

1. Primary Outcome: Delis-Kaplan Executive Function System Verbal Fluency
Description: Number of words per category in one minute
Time Frame: 5-15 minutes following stimulation frequency setting change.
Measure: Mean (Standard Error); unit: Words per minute
Arm/Group | STN DBS Off | STN DBS 10Hz | STN DBS 130Hz
Number analyzed (Participants) | 12 | 12 | 12
Words per minute
  Letter | 12.75 (1.7) | 13.25 (1.54) | 13.58 (1.54)
  Nonepisodic | 13.83 (1.36) | 11.33 (2.93) | 11.83 (1.11)
  Episodic | 17.17 (1.56) | 18.00 (1.47) | 15.46 (1.47)
  Category Switching | 14 (1.76) | 25.00 (5.23) | 13.17 (0.94)

2. Primary Outcome: Delis-Kaplan Executive Function System Color Word Interference Task
Description: Time to completion of a color-word interference task
Time Frame: 5-15 minutes following stimulation frequency setting change.
Measure: Mean (Standard Error); unit: Seconds
Arm/Group | STN DBS Off | STN DBS 10Hz | STN DBS 130Hz
Number analyzed (Participants) | 12 | 12 | 12
Seconds
  Color reading | 33.83 (2.68) | 35.00 (2.51) | 34.33 (6.61)
  Word reading | 24.58 (1.96) | 24.75 (1.74) | 24.17 (5.62)
  Color-word interference | 67.92 (4.58) | 70.00 (6.84) | 67.92 (10.54)
  Color-word switching | 72.42 (7.17) | 74.25 (7.74) | 70.25 (18.98)

3. Primary Outcome: Random Number Generation
Description: Listing of 100 numbers at 1 Hz in a random order.
  Evan's RNG: a measure of disproportion with which one number follows another in a sequence. Scores range from 0 (equal proportion of sequence pairs) to 1 (maximum disproportion of sequence pairs). A higher score indicates a lower randomness and poorer exective function.
  Count score 1: a measure of propensity to count in steps of 1. The length of each sequence with steps of 1 is squared. The total of these is summed. Scores range from 0 (no sequences with steps of 1) to 100000 (all sequences with steps of 1). A higher score indicates lower randomness and poorer exective function.
  Count score 2: a measure of propensity to count in steps of 2. The length of each sequence with steps of 2 is squared. The total of these is summed. Scores range from 0 (no sequences with steps of 2) to 100000 (all sequences with steps of 2). A higher score indicates lower randomness and poorer exective function.
  Evan's RNG, count score 1 and cou
Time Frame: 5-15 minutes following stimulation frequency setting change.
Measure: Mean (Standard Error); unit: Index
Arm/Group | STN DBS Off | STN DBS 10Hz | STN DBS 130Hz
Number analyzed (Participants) | 12 | 12 | 12
Index
  Evan's RNG | 0.35 (0.02) | 0.35 (0.02) | 0.37 (0.01)
  Count score 1 | -3.10 (0.41) | -3.21 (0.38) | -2.90 (0.34)
  Count score 2 | -3.27 (0.29) | -2.65 (0.40) | -2.32 (0.25)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the entire duration of the study, which lasted between 3 and 4 hours. Patients were assessed at a mean of 21.4 (range 7-52) months following bilateral STN DBS insertion.
Arm/Group | STN DBS Off | STN DBS 10Hz | STN DBS 130Hz
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12

LIMITATIONS AND CAVEATS:
Our study did not control for motor state during testing. Our sample population was not fully representative of the worldwide population of patients with PD.

Our study was not designed nor powered to investigate inter-subject differences such as age, time from DBS implantation, education, first language, or motor function.

Unknown is the adequacy of a 5-min period of stimulation prior to each round of neuropsychological testing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-03): https://cdn.clinicaltrials.gov/large-docs/65/NCT04383665/Prot_SAP_000.pdf
  • Informed Consent Form (2019-10-25): https://cdn.clinicaltrials.gov/large-docs/65/NCT04383665/ICF_001.pdf